CLINICAL TRIAL: NCT01381354
Title: Nutrition, Neuromuscular Electrical Stimulation (NMES) and Secondary Progressive Multiple Sclerosis (SPMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Direct MS Canada (Unknown); DJO Incorporated (Industry); Pinnaclife Inc. (Industry); TZ Press, LLC (Unknown)
Responsible Party: Principal Investigator, Terry L. Wahls, Clinical Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200911781
Record Dates: First submitted 2011-05-26; First posted 2011-06-27 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis, primary progressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Diet, Paleolithic; Diet, Gluten-Free; Fatty Acids, Omega-3; Magnesium; Niacinamide; Taurine; Creatine; Thiamine; Riboflavin; Acetylcysteine; Thioctic Acid; Acetylcarnitine; 5-methyltetrahydrofolate; Ubiquinone; Meditation; Educational Status; Coconut Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined intervention (Experimental): Combination intervention consisting of the following: structured modified paleolithic diet, Progressive Exercise, Neuromuscular Electrical Stimulation designed to facilitate the adoption of multiple therapeutic lifestyle behaviors associated with superior health outcomes.
  Interventions: Other: Progressive exercise; Device: Neuromuscular electrical stimulation delivered using the electrical therapy device EMPI 300 PV; Other: Modified paleolithic diet; Dietary Supplement: Omega 3 fatty acids; Dietary Supplement: Full Spectrum vitamin; Dietary Supplement: Essential - hydroxytyrosol; Dietary Supplement: Maltodextrin fiber supplement; Dietary Supplement: Mineral boost (magnesium); Dietary Supplement: Niacinamide; Dietary Supplement: Methyl B12; Dietary Supplement: Taurine; Dietary Supplement: creatine; Dietary Supplement: thiamine; Dietary Supplement: riboflavin; Dietary Supplement: N acetylcysteine; Dietary Supplement: alpha lipoic acid; Dietary Supplement: L acetyl carnitine; Dietary Supplement: methyl folate; Dietary Supplement: coenzyme Q; Behavioral: meditation; Behavioral: self massage; Behavioral: learning; Dietary Supplement: Coconut oil

INTERVENTIONS:
Other: Progressive exercise — Progressive strengthening exercises designed to improve core muscles and muscles of ambulation.
Device: Neuromuscular electrical stimulation delivered using the electrical therapy device EMPI 300 PV — Neuromuscular electrical stimulation to train core muscles and ambulation muscles. Device is Empi 300 manufactured by DJO Inc.
  Other Names: NMES, electrical therapy
Other: Modified paleolithic diet — Diet based upon a Paleolithic diet and structured to increase the consumption of greens, sulfur rich vegetables, bright colors, seaweed and omega 3 fatty acid rich foods.
  Other Names: Wahls Diet, Paleolithic Diet, Gluten-free, Dairy-free.
Dietary Supplement: Omega 3 fatty acids — 4 grams daily by mouth.
  Other Names: Pinnaclife Omega 3 fatty acids
Dietary Supplement: Full Spectrum vitamin — Two capsules daily.
  Other Names: Pinnaclife
Dietary Supplement: Essential - hydroxytyrosol — Two capsules twice daily.
  Other Names: Pinnaclife Essential
Dietary Supplement: Maltodextrin fiber supplement — One scoop daily.
  Other Names: Pinnaclife Cleanse
Dietary Supplement: Mineral boost (magnesium) — Two capsules daily
  Other Names: Pinnaclife Mineral Boost.
Dietary Supplement: Niacinamide — 500 mg daily
Dietary Supplement: Methyl B12 — Methyl B12 1000 mcg daily
Dietary Supplement: Taurine — one gram daily
Dietary Supplement: creatine — one teaspoon daily
Dietary Supplement: thiamine — 100 mg daily
Dietary Supplement: riboflavin — 200 mg daily
Dietary Supplement: N acetylcysteine — 1 gram daily
Dietary Supplement: alpha lipoic acid — 300 mg twice daily
Dietary Supplement: L acetyl carnitine — 500 mg twice daily
Dietary Supplement: methyl folate — 1000 mcg one pill four times a week
Dietary Supplement: coenzyme Q — 100 mg daily
Behavioral: meditation — meditation 15 minutes daily
Behavioral: self massage — self massage of hands, feet, ears 15 minutes daily
Behavioral: learning — completing puzzles or learning 15 minutes daily
Dietary Supplement: Coconut oil — If excessive weight loss occurs, the subject will add 1-2 tablespoons of coconut oil daily to smoothies or foods eaten.
  Other Names: Extra virgin cold press coconut oil

SUMMARY:
The study will use a multimodal therapeutic lifestyle intervention consisting of a study diet, stressing more vegetables and fruit, elimination of foods at greatest risk for food allergy, meditation, self massage, progressive exercise and neuromuscular electrical stimulation for rehabilitation of gait and fatigue disability in the setting of secondary and primary progressive multiple sclerosis with gait disability.

DETAILED DESCRIPTION:
Restoration of function is very rare in individuals with MS who have experienced gradual worsening in the absence of acute MS symptoms (relapses) and partial or complete recovery of those acute symptoms (remissions).

A recent case report of a patient with secondary progressive MS documented a transition from scooter dependence to mild gait disability following the initiation of electrotherapy in the form of neuromuscular electrical stimulation and nutritional interventions aimed increasing the nutrient density and decreasing the risk of food sensitivity and food allergies. Multiple studies of neuromuscular electrical stimulation in athletes, cerebral palsy and stroke patients have demonstrated gains in strength and coordination. Multiple authors have reported that antioxidants, essential amino acids and micronutrient rich diets are neuroprotective. It is likely that the combination of the intensive nutrition and the electrotherapy contributed to the marked gains in improvement. However in the absence of an additional case report the strength of the association remains unknown.

The intent of this study is to replicate the interventions from the case report as closely as possible.

Our primary objective is to measure how many and how completely subjects implement 1) the nutritional interventions, 2) the home exercise program intervention, and 3) the electrotherapy intervention and if the improve improved nutrition and exercise are associated with improved function. To assess improvements in function will measure 1) the change in nutritional status as reported in food frequency surveys, 24 hr dietary recalls, 2) change in neurocognitive testing and behaviors, 3) change in self-reported function and disability scales, 4) change in gait and 5) change in medications doses or classes for MS related symptoms.

Subjects will be followed for three years. After the first year, subjects will not receive intensive support from the study team. The subjects return at months 18, 24 and 36 to assess adherence with study interventions, function and quality of life. Nutrition intake is assessed again at 24 and 36 months.

To assess for safety we will assess safety labs (kidney and liver function tests) and changes in weight, and self reported side effects questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Secondary or primary progressive multiple sclerosis
* Some level of gait disability
* Tolerance for test electrical therapy session
* Successful completion of two week Run-IN phase completing the daily logs -
* Demonstrating > 80% compliance with dietary and behavioral interventions

Exclusion Criteria:

* Antiplatelet or blood thinning medication
* Cognitive disability or psychiatric disorder making compliance with study interventions difficult
* Implanted electronic medical device
* Change in medication in the prior three months
* Active cancer treatment (skin basal cell or squamous cancer is not an exclusion criteria)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Fatigue severity scale | Baseline, 3 M, 6M, 9M,12 M
  Self reported fatigue severity scale, (agreement with 9 questions describing impact of fatigue on daily activities)

SECONDARY OUTCOMES:
25 foot walk | baseline, 3M, 6M, 9M, 12M, 18M, 24M 36M
  Average walking speed calculated from 25 foot walk. Distance (feet)walked divided by time in seconds.
  Step and stride length, step and stride duration.
Short Form 36 | baseline, 3M, 6M, 9M, 12M, 18M, 24M, 36 M
  Self reported function in multiple domains.
Mood scales | Baseline, 3 M, 6M, 9M, 12M
  Beck depression index, Beck anxiety index
Cognitive Scales | baseline, 3 M, 6M, 9M, 12 M
  Cognitive stability index or cognitive stability test, subscales of Dkef, Wtar, Wais III.
Medical Symptoms Questionnaire | baseline, 1 M, 2M, 3M, 4M, 5M, 6M, 7M, 8M, 9M, 10 M, 11M, 12M, 18M, 24M, 36M
  Detailed review of systems which is scored 0 to 4 for each item.
Side effects log | Baseline, 1M, 2M, 3M, 4M, 5M, 6M, 7M, 8M, 9M, 10 M, 11M, 12M
  Questions about potential side effects from vitamin, supplements and diet, questions about potential side effects from NMES, and questions about potential side effects from exercise.
MS Function | Baseline, 3 M, 6M, 9M, 12M, 18M, 24M, 36M
  Self reported disability scales (from North American Research committee on Multiple Sclerosis)
Multiple Sclerosis Spasticity Scale-88 | Baseline, 3M, 6M,9M and 12M, 18M, 24M, 36M
  88 Questions about the impact of spasticity on various activities of daily living
Daily log | Baseline, 1M, 2M, 3M, 4M, 5M, 6M, 7M, 8M, 9M, 10 M, 11M, 12M
  Daily reports of foods consumed, exercises and activities completed.
Vitamin log | Baseline, 1M, 2M, 3M, 4M, 5M, 6M, 7M, 8M, 9M, 10 M, 11M, 12M
  Log of vitamins supplement bottles date opened, date emptied, pill size, number of pills in bottle.
Medical examination | Baseline, 12 M
  Medical examination
Neurological examination | Baseline and 12 M
  Neurological examination
Exposure history form | Baseline
  History of exposures to chemicals.
Health questions | Baseline
  health questions about chronic disease states
Menses and pregnancy risk | Baseline, 3M, 6M, 9M, 12M
  Questions about menses and potential for pregnancy
Medication audit | Baseline, 12 M
  Medications
Functional diagnoses | Baseline
  Questions about past medical history
Manual motor testing | Baseline, 3M, 6M, 9M, 12M
  Manual motor testing of arms, legs and core muscle groups.
Berg Balance | baseline, 3M, 6M, 9M, 12M
  Tests of balance which are progressively more challenging.
Modified Ashworth | baseline, 3M, 6M, 9M, 12M
  Test of spasticity by physical examination.
Circumference | baseline, 3M, 6M, 9M, 12M
  Circ. of waist, hips, R and+ L calf and R. and L. thigh.
Peak flow | baseline, 3M, 6M, 9M, 12M
  Peak expiratory flow rate.
Number of falls in prior two months | Baseline, 3M, 6M, 9M,12M, 18M, 24M, 36M
  Self reported number of falls and associated factors contributing to fall and severity of fall related injuries.
Dietary compliance | Baseline, 6 month and 12 month, 36 month
  Assessments, self report, Harvard Food Frequency (baseline, 12 month), 24 hour dietary recalls (6M)
Blood pressure | baseline, 3M, 6M, 9M, 12M
  blood pressure
Waist/ Hip ratio | baseline, 3M, 6M, 9M, 12M
  circumference of waist over the circumference of hip
MS quality of life- 54 | Baseline and months 3,6,9,12,18,24,and 36
  Quality of life questionnaires asking about various aspects of daily life.
Blood Biomarkers | Baseline, 12 months
  Blood biomarkers of inflammation, and nutritional status.
Change in functional and structural brain Magnetic Resonance Imaging (MRI) measures | Between 1 and 12 month post intervention
  Following sequences:
  T1 weighted - Pre Gadolinium T1 weighted -Post Gadolinium T2 weighted FLAIR functional MRI during cognitive task Resting state functional MRI Diffusion Tensor Imaging
Fatigue severity scale | 18 M, 24 M, 36 M
  Self reported fatigue severity scale, (agreement with 9 questions describing impact of fatigue on daily activities)
Get up and go test time | Baseline, 3M, 6M, 9M, 12M, 18M, 24M, 36M
  Total time to get up from chair, walk 10 feet and come back and sit down on the chair.
  Step and stride length, step and stride duration and double support time.
Change in weight and Body mass index (BMI) | Baseline, 3M, 6M, 9M, 12M, 18M, 24M, 36M
  weight measured in Kg Body mass index (BMI)
Blood safety biomarkers | Baseline, 1M, 3M, 6M, 9M, 12M, 18M, 24M, 36M
  Kidney and liver function tests and complete blood count
9 hole peg board test | Baseline, 3M, 6M, 9M,12M, 18M, 24M, 36M
  Time to put 9 pegs in holes and take them out.
Paced auditory serial addition task (PASAT) | Baseline, 3M, 6M,9M,12M, 18M,24M,36M
  Addition of two consecutive numbers during a series of numbers heard by subject.
Veteran specific activity questionnaire | Baseline, 3M, 6M, 9M, 12M, 18M,24M,36M
  Questions about the maximum physical activity level.
Form 38- Daily life | 12M, 18M, 24M, 36M
  Questions about stressful life events.
Urine toxicology | Baseline and 12 M
  24 hours urine collection and measurement of heavy metals.
Stool microbial profile | Baseline and 12M
  DNA probe for bacteria, parasites and yeast DNA.
Harvard food frequency questionnaire and 24 hour food recalls | Baseline, 12M, 24M and 36M
  Questions regarding food intake and frequency of type of food consumed in last one year.
  Phone interview asking about food consumed in last 24 hours.
Bio impedance analysis | Baseline, 12M, 24M and 36M
  Test to analyze body composition.
Exercise and electrical stimulation daily log | Daily baseline through 12M, 14 day-logs before/after 18M, 24M and 36M
  Record of exercise, use of electrical stimulation on muscles and physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Iowa/ VA Iowa City VA Medical Center, Iowa City, Iowa, United States

REFERENCES:
- [Background] Wahls TL, Reese D, Kaplan D, Darling WG. Rehabilitation with neuromuscular electrical stimulation leads to functional gains in ambulation in patients with secondary progressive and primary progressive multiple sclerosis: a case series report. J Altern Complement Med. 2010 Dec;16(12):1343-9. doi: 10.1089/acm.2010.0080. PMID 21138391
- [Background] Reese D, Shivapour ET, Wahls TL, Dudley-Javoroski SD, Shields R. Neuromuscular electrical stimulation and dietary interventions to reduce oxidative stress in a secondary progressive multiple sclerosis patient leads to marked gains in function: a case report. Cases J. 2009 Aug 10;2:7601. doi: 10.4076/1757-1626-2-7601. PMID 19918474